CLINICAL TRIAL: NCT00233870
Title: Special Survey in Long-Term Use of Fabrazyme
Brief Title: A Long Term Safety and Efficacy Study of Fabrazyme Replacement Therapy in Japanese Patients With Fabry Disease.
Status: Completed | Type: Observational
Sponsor: Genzyme, a Sanofi Company (Industry)
Responsible Party: Sponsor
Organization: Sanofi (Industry)
Other Study IDs: AGAL03004
Record Dates: First submitted 2005-10-05; First posted 2005-10-06 (Estimated); Last update posted 2015-05-08 (Estimated); Status verified 2015-05

CONDITIONS: Fabry Disease
MeSH Terms: conditions — Fabry Disease | interventions — agalsidase beta

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

INTERVENTIONS:
Drug: Agalsidase beta (recombinant form) — agalsidase beta 1.0 mg/kg body weight infused every 2 weeks as an intravenous infusion
  Other Names: Fabrazyme

SUMMARY:
The purpose of this survey is to identify any concerns regarding the following efficacy and safety-related issues in clinical practice with the new drugs "Fabrazyme for intravenous infusion 5mg" and "Fabrazyme for intravenous infusion 35mg" and to confirm the safety of these products in long-term use in the clinical setting.

1. New adverse drug reactions (ADRs) that cannot be predicted from the Precautions (in particular, clinically significant ADRs)
2. The incidence of ADRs under the actual conditions of use of the drug
3. Causal factors that might potentially affect safety
4. Efficacy evaluation in long-term use

This survey will be conducted in accordance with the approval condition established for Fabrazyme:

"To conduct a special surveillance of Efficacy and Safety in long term treatment and Pediatric with the drug."

DETAILED DESCRIPTION:
Medical institutions or physicians will be asked to periodically complete the survey forms for all patients registered. Survey forms include baseline information available, and then data collected every 6 months, as available including: demographic information, concomitant medications/therapy, treatment record, ECG, Echocardiogram, computed tomography scan / magnetic resonance imaging (CT/MRI), Fabry symptoms, labs, functional disorder, blood concentration of GL-3, and anti-agalsidase beta antibody test (IgE testing) to survey whether the productions of antibodies to agalsidase beta is a causal factor of treatment-related reactions.

The survey period shall be approximately 7 years from June 1, 2004 during which survey shall be undertaken as follows:

* The observation period for each patient shall range from 1 to about 7 years after starting treatment
* Registration period: June 1, 2004 to March 31, 2010
* Survey period: June 1, 2004 to March 31, 2011

In institutions for which retrospective surveys are feasible, the survey period will trace back to the date of approval (January 29, 2004), as far as possible.

ELIGIBILITY:
Inclusion Criteria:

* Patients in Japan with the indication of "Fabry Disease" and for whom the usual dosage and administration is 1mg of agalsidase beta (recombinant) per 1 kg body weight each time, administered by intravenous infusion every 2 weeks
* Because the efficacy evaluation of enzyme replacement therapy with Fabrazyme [agalsidase beta (recombinant form)] will require the comparison of findings before and after the start of enzyme replacement therapy, the efficacy evaluation set will be defined as including patients using Fabrazyme [agalsidase beta (recombinant form)] for the first time in the post-marketing setting and those for whom it is possible to obtain retrospective data for before the start of enzyme replacement therapy.

Exclusion Criteria:

* Patients registered in the post-marketing trials during the post-marketing clinical trial period.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Japanese patients with Fabry Disease
Sampling Method: Non-Probability Sample
Enrollment: 405 (Actual)
Dates: Start 2004-06; Primary Completion 2011-03 (Actual); Study Completion 2011-03 (Actual)

PRIMARY OUTCOMES:
Change in blood GL-3 level | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Genzyme, a Sanofi Company
Locations (1):
- Tohoku University Hospital, Sendai, Japan

REFERENCES:
- [Derived] Lee CS, Tsurumi M, Eto Y. Safety and tolerability of agalsidase beta infusions shorter than 90 min in patients with Fabry disease: post-hoc analysis of a Japanese post-marketing study. Orphanet J Rare Dis. 2023 Jul 24;18(1):209. doi: 10.1186/s13023-023-02803-5. PMID 37488580
- [Derived] Tsurumi M, Suzuki S, Hokugo J, Ueda K. Long-term safety and efficacy of agalsidase beta in Japanese patients with Fabry disease: aggregate data from two post-authorization safety studies. Expert Opin Drug Saf. 2021 May;20(5):589-601. doi: 10.1080/14740338.2021.1891221. Epub 2021 Mar 10. PMID 33599146